CLINICAL TRIAL: NCT04455204
Title: Implication of Adipokines, Inflammation, Insulin Resistance and Endothelial Dysfunction in the Pathogenesis of Preeclampsia and in Pregnancy Related Complications
Brief Title: Adipokines, Inflammation, Insulin Resistance and Endothelial Dysfunction in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Dr. Tarek Mohamed Mostafa, Associate Professor, Tanta University
Other Study IDs: CP0002
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Pre-Eclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-pregnant women (group 1): 20 non-pregnant women who serve as a control group (group 1)
  Interventions: Diagnostic Test: Serum asymmetteric dimethyl arginine; Diagnostic Test: serum lipid profiles; Diagnostic Test: Serum vaspin; Diagnostic Test: Serum resistin
- pregnant women (group 2): 20 pregnant women with normal pregnancy at their third trimesters (group 2)
  Interventions: Diagnostic Test: Serum asymmetteric dimethyl arginine; Diagnostic Test: serum lipid profiles; Diagnostic Test: Serum vaspin; Diagnostic Test: Serum resistin
- pregnant women with Preeclampsia (group 3): 20 pregnant women with Preeclampsia in their third trimester (group 3) will be screened to fit the inclusion and exclusion criteria.
  Interventions: Diagnostic Test: Serum asymmetteric dimethyl arginine; Diagnostic Test: serum lipid profiles; Diagnostic Test: Serum vaspin; Diagnostic Test: Serum resistin

INTERVENTIONS:
Diagnostic Test: Serum asymmetteric dimethyl arginine — Serum asymmetteric dimethyl arginine (ADMA) will be done using Enzyme-Linked Immunosorbent Assay
  Other Names: ADMA
Diagnostic Test: serum lipid profiles — serum lipid profiles including triglycerides (TG), total cholesterol and high-density lipoprotein cholesterol (HDL-C) which will be measured by enzymatic colorimetric method) using commercial kits
  Other Names: Lipids
Diagnostic Test: Serum vaspin — vaspin concentrations will be assayed using commercially available ELISA kits
Diagnostic Test: Serum resistin — resistin concentrations will be assayed using commercially available ELISA kits

SUMMARY:
The aim of the present study is to evaluate the implication of adipokines, inflammation, insulin resistance and endothelial dysfunction in the pathogenesis of preeclampsia and in pregnancy related complications.

DETAILED DESCRIPTION:
This observational parallel study will be conducted on pregnant women with normal pregnancy, pregnant women with Preeclampsia, and on healthy non-pregnant women. All participants will be recruited from the Outpatient Clinic of Obstetrics and Gynecology Department at Menoufia University Hospital (Shebin El-Kom, Egypt). The study will be approved by the Research Ethics Committee of Menoufia University and all the involved subjects will give their written informed consent.

This study will involve a total number of 60 women who will be further classified into: 20 non-pregnant women who serve as the control group (group 1), 20 pregnant women with normal pregnancy at their third trimesters (group 2) and 20 pregnant women with Preeclampsia at their third trimester (group 3) will be screened to fit the inclusion and exclusion criteria. The pregnant women will be assessed in their third trimesters and further re-evaluated 4 weeks after delivery. The gestational ages will be determined conventionally and re-affirmed by ultrasonographic measurement.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with normal pregnancy (n=20)
* Pregnant women with Preeclampsia (n=20) at their third trimesters of pregnancy will be included in the study. Preeclampsia will be defined and diagnosed by constant elevation in blood pressure greater than 140/90 mmHg and by the presence of proteinuria above 300 mg /24 hour with the absence of both urinary tract infection and previous history of hypertension.
* Apparently healthy non-pregnant females (n=20) will be included in this study also.

Exclusion Criteria:

* Women with risk factors for oxidative stress such as smokers and
* Those with a medical history of diabetes mellitus (DM) and Tuberculosis (T.B).
* Women with a history of hypertension, familial hyperlipidemia, liver diseases, inflammatory diseases, and renal impairment.
* Non-pregnant women on hormonal therapy or hormonal contraceptives.

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: total number of 60 women who will be further classified into: 20 non-pregnant women who serve as control group (group 1), 20 pregnant women with normal pregnancy at their third trimesters (group 2) and 20 pregnant women with Preeclampsia at their third trimester (group 3) will be screened to fit the inclusion and exclusion criteria. The pregnant women will be assessed in their third trimesters and further re-evaluated 4 weeks after delivery. The gestational ages will be determined conventionally and re-affirmed by ultrasonographic measurement.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Interleukin 18 | Nine months
  IL-18 will be carried out using Enzyme-Linked Immunosorbent Assay
Vaspin level | Nine months
  Serum vaspin concentrations will be assayed using commercially available ELISA kits
resistin level | Nine months
  Serum resistin concentrations will be assayed using commercially available ELISA kits
Malondialdehyde level | Nine Months
  MDA will be measured spectrophotometrically
Serum asymmetteric dimethyl arginine (ADMA) | Nine Months
  Serum asymmetteric dimethyl arginine (ADMA) will be done using Enzyme-Linked Immunosorbent Assay
insulin resistance (IR) | Nine Months
  insulin resistance (IR) using the HOMA-IR index [18], which is defined as fasting insulin (μIU/ml) times fasting glucose (mmol/l) divided by 22.5 or divided by 405 if fasting blood glucose is expressed in mass units (mg/dl).

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Mostafa, Ass. Prof., Study Director — Tanta University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jia X, Wang S, Ma N, Li X, Guo L, Liu X, Dong T, Liu Y, Lu Q. Comparative analysis of vaspin in pregnant women with and without gestational diabetes mellitus and healthy non-pregnant women. Endocrine. 2015 Mar;48(2):533-40. doi: 10.1007/s12020-014-0318-7. Epub 2014 Jun 15. PMID 24929806
- [Background] Jahromi AS, Shojaei M, Ghobadifar MA. Insulin resistance and serum levels of interleukin-17 and interleukin-18 in normal pregnancy. Immune Netw. 2014 Jun;14(3):149-55. doi: 10.4110/in.2014.14.3.149. Epub 2014 Jun 19. PMID 24999311